CLINICAL TRIAL: NCT05719116
Title: A Combined Aerobic and Resistance Training Program for Adults With Psychotic Disorders
Acronym: TREPP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Solli Distriktspsykiatriske Senter (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-17695
Record Dates: First submitted 2022-11-23; First posted 2023-02-08 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: As the main aim of the study is to investigate feasibility, no randomisation is done at this stage. The participants with psychotic disorder will be compared with participants with a psychiatric disorder (but no psychotic disorder).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical exercise for participants with psychotic disorder (Experimental): Participants with a psychotic disorder will exercise in a group supervised by a physiotherapist for 16 weeks, three times a week.
  Interventions: Behavioral: Physical exercise
- Physical exercise for participants with psychiatric disorder, but not psychotic disorder (Active Comparator): Participants with a psychiatric disorder will exercise in a group supervised by a physiotherapist for 16 weeks, three times a week.
  Interventions: Behavioral: Physical exercise

INTERVENTIONS:
Behavioral: Physical exercise — The physical exercise will be aerobic and strength training. The sessions will last app. 1 hour.

SUMMARY:
The study is a feasibility study of a combined high intensity aerobic and strenght exercise program for persons with psychotic disorders. The feasibility of the protocol will be investigated, in addition to the participants subjective experience with the participation.

DETAILED DESCRIPTION:
The aim of this study is to investigate the feasibility of a 16 week physical exercise intervention combining strenght and aerobic training in group for patients with psychotic disorders. In addition, the feasibility of the test protocol and participants subjective experience with the intervention will be investigated.

Research shows positive effects of physical exercise for patients with psychotic disorders regarding maximal aerob training, maximal muscle strength, physical, cognitive and social functioning, and symptom levels. Effects and the degree of feasibility of physical exercise for patients with psychotic disorders are amplified by regarding their preferences and needs, and if they experience support and guidance during the intervention. Earlier studies have focused mostly on either strength og endurance training, or combined interventions of moderate intensity. We now want to investigate the feasibility of an invidually adjusted combined program of high intensity.

After the intervention, participants will be interviewed about their experience with participating.

ELIGIBILITY:
Participants with psychotic disorder:

Inclusion Criteria:

* Signed informed consent
* Diagnosed with psychotic disorder
* Physically able to participate in physical exercise
* Is a patient at Solli DPS
* Motivated for participating in physical exercise

Exclusion Criteria:

* Physical conditions precluding the participant from the physical testing/training
* Mental state that hinders participation, such as ongoing suicidality, substance abuse or brain organic disorder

Participants with psychiatric disorder, but no psychotic disorder:

Inclusion Criteria:

* Signed informed consent
* Diagnosed with psychiatric disorder, but not a psychotic disorder
* Physically able to participate in physical exercise
* Is a patient at Solli DPS
* Motivated for participating in physical exercise

Exclusion Criteria:

* Physical conditions precluding the participant from the physical testing/training
* Mental state that hinders participation, such as ongoing suicidality, substance abuse or brain organic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention program | After 16 weeks of intervention
  How many participants completed the physical training intervention.

SECONDARY OUTCOMES:
Aerobic capasity: Ekblom Bak submaximal ergometer cycle test | At week 0 and 16
  Estimating Vo2max
Aerobic capasity: 4 x 4 interval for estimating VO2max | At week 0 and 16
  Standarised 4x4 interval training for estimating VO2max with the smartphone app My Workout GO
Strength: 1 RM test of bench press | At week 0 and 16
  Maximal test of strenght of upper body
Strenght: 1 RM test of squat | At week 0 and 16
  Maximal test of lower body musculature
Psychotic symptoms: The Positive and Negative Syndrome Scale | At week 0 and 16
  For the participants with psychotic disorders only. A measure of positive and negative psychotic symptoms. Each item is scored on a scale from 1-7 with a higher score indicating higher symptom level.
Depression symptoms: The Calgary Depression Scale for Schizophrenia | At week 0 and 16
  A measure of depressive symptoms. Each item is scored on a scale from 0-3 with a higher score indicating higher symptom level.
Anxiety symptoms: GAD-7 | At week 0 and 16
  A measure of anxiety symptoms. This is a 7-item self-report questionnaire where participants rate on a scale from 0 (not at all sure) to 3 (nearly every day). A higher score indicates greater symptom severity.
Quality of life: SF-12 | At week 0 and 16
  A measure of health related quality of life. The items is scored after variying categories such as "yes" and "no", and "How much time during the past 4 weeks...".

OTHER OUTCOMES:
In depth interview | After 16 weeks of intervention
  A semi structured interview for asking the participants about their experience with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Sirevåg, Principal Investigator — Solli DPS
Locations (1):
- Solli DPS, Bergen, Nesttun, Norway

IPD SHARING:
Plan to Share IPD: Yes
We plan to publish our results in peer-reviewed journals.
Supporting Information: Study Protocol, SAP
Time Frame: We plan to publish the study protocol. The statistical analysis plan will be available in published articles.
Access Criteria: After data collection has been completed, data can be available upon reasonable request.